CLINICAL TRIAL: NCT03893981
Title: Comparison of the Effect of Strengthening Exercises Versus Proprioception and Balance Exercises in the Treatment of Knee Osteoarthritis
Brief Title: Strengthening Exercises Versus Proprioception and Balance Exercises in the Treatment of Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Gamze Kus, Principal Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 99984023-302.99
Record Dates: First submitted 2019-03-07; First posted 2019-03-28 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Osteo Arthritis Knee; Pain
Keywords: Rehabilitation; Pain; Functionality; Proprioception
MeSH Terms: conditions — Pain | interventions — Proprioception; Resistance Training

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proprioception and Balance Training (Experimental): Proprioception and Balance Program
  Interventions: Other: Proprioception and Balance Program
- Strengthening Training (Experimental): Strengthening Program
  Interventions: Other: Strengthening Program

INTERVENTIONS:
Other: Proprioception and Balance Program — Balance Trainer device and playing ball in tandem position for using to improve balance, vibration and reposition exercises for using to improve proprioception. Progressive of training will increase after each 2 weeks.Patients will be taken to the treatment program 3 days in a week for 8 weeks.
  Arms: Proprioception and Balance Training
Other: Strengthening Program — Exercises which include open and closed kinetic chain exercise will be applied to strength knee and hip muscle. Progressive of training will increase after each 2 weeks. Patients will be taken to the treatment program 3 days in a week for 8 weeks.
  Arms: Strengthening Training

SUMMARY:
The aim of the study is to investigate and compare the effect of balance and proprioception exercises with strengthening exercises on muscle strength, pain, proprioception, function and quality of life in knee osteoarthritis patients.

DETAILED DESCRIPTION:
Damage or loss of mechanoreceptors in osteoarthritis patients affects balance and proprioception. There are studies showing that proprioceptive deficit is associated with the onset and progression of knee osteoarthritis leading to pain and disability. Because the proprioception provides a sense of power generation and allows the power output to be better regulated. When the literature is examined, studies investigating the effects of proprioception and balance exercises on muscle strength, function and pain are limited.

In our study patients will be randomly divided into two groups: Group I (Proprioception and Balance) and Group II (muscle strengthening exercises). While Group I will be applied Proprioception and Balance training exercises, Group II will be applied closed and open kinetic strengthening exercises. Two group will perform exercise 3 times a week during 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have a diagnosis of knee Osteoarthritis according to the American Society of Rheumatology (ACR) criteria,
* Between 45 to 75 years of age
* Can read and write in Turkish language

Exclusion Criteria:

* Active synovitis
* Taking any physical therapy section in the last 6 months
* Have a neurological problems that affect walking
* Have an arthritis problem in the ankle and hip joint
* Have a history of lower extremity surgery
* Intraarticular steroid injection in the last 6 months
* Use psychoactive drug
* Have a severe defect of vision and hearing, speech disorders
* Vestibular dysfunction

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2020-08-11 (Actual); Study Completion 2020-08-11 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Arthritis Index (WOMAC) | WOMAC will be filled first time at baseline and second time after 4 weeks and third time after 8 weeks rehabilitation program . After treatment "change" will be assessed
  The WOMAC is widely used self-administered health status measure used in assessing pain, stiffness and function in patients with OA of the knee or hip. The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
  The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) | Evaluation will perform first time at baseline and second time after 4 weeks and third time after 8 weeks rehabilitation program.
  The Visual Analog Scale (VAS) is a 10 cm line with anchor statements on the left (no pain) and on the right (extreme pain). The patient is asked to place a vertical mark on the scale to indicate the level of intensity of his or her pain.
Pressure Algometer | Evaluation will perform first time at baseline and second time after 4 weeks and third time after 8 weeks rehabilitation program.
  Pressure algometry is one of a number of outcome measures that manual therapy practitioners are able to use in both clinical and research settings. The pressure algometer is used to determine the pressure pain threshold of specific muscle and bone locations.
Hand-Held Dynamometer | Evaluation will perform first time at baseline and second time after 4 weeks and third time after 8 weeks rehabilitation program.
  Handheld dynamometers are one of the most objective and consistent tools to use when muscle testing. It is an ergonomic hand-held device for objectively quantifying muscle strength.
Isokinetic Dynamometer for measuring position sense | Evaluation will perform first time at baseline and second time after 4 weeks and third time after 8 weeks rehabilitation program.
  Isokinetic dynamometer is a well known device to measure active and passive JPS and also provides target angle result without any researcher bias/It has shown good reliability and validity for measuring position sense.
Short Form-36 | Evaluation will perform first time at baseline and second time after 4 weeks and third time after 8 weeks rehabilitation program.
  The Short Form (36) Health Survey is a 36-item, patient-reported survey of health related quality of life. The RAND 36-Item Health Survey taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health.
Global Rating of Change Scale | Evaluation will perform first time at baseline and second time after 4 weeks and third time after 8 weeks rehabilitation program.
  Global rating of change (GRC) scales are very commonly used in clinical research, particularly in the musculo-skeletal area These scales are designed to quantify a patient's improvement or deterioration over time, usually either to determine the effect of an intervention or to chart the clinical course of a condition. Global Rating of Change Scale will be used to evaluate patients' satisfaction from treatment.
Aggregated Locomotor Function (ALF) Score | Evaluation will perform first time at baseline and second time after 4 weeks and third time after 8 weeks rehabilitation program.
  The aggregated locomotor function (ALF) score, a simple measure of observed locomotor function, using timed walking, stairs and transfers, was developed and evaluated for intra-tester reliability, criterion-related validity and responsiveness in a sample of patients with knee osteoarthritis.
Digital Goniometer | Evaluation will perform first time at baseline and second time after 4 weeks and third time after 8 weeks rehabilitation program.
  Digital Goniometer is a tool used most commonly for evaluating joint ROM in the clinical settings. Also it is a simple alternative for global use.
Timed Up and Go (TUG) Test | Evaluation will perform first time at baseline and second time after 4 weeks and third time after 8 weeks rehabilitation program.
  Timed Up and Go (TUG) Test will be used clinical performance-based measure of lower extremity function, mobility and fall risk.
Tandem and Stand on One Leg | Evaluation will perform first time at baseline and second time after 4 weeks and third time after 8 weeks rehabilitation program.
  Tandem and Stand on One Leg will ve used to assesment of static balance of patients

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Kuş, MsC, Principal Investigator — Istanbul University
Locations (1):
- Istanbul University-Cerrahpasa, Faculty Of Health Sciences, Istanbul, Bakirkoy, Turkey (Türkiye)